CLINICAL TRIAL: NCT00875472
Title: Social Influences on Adolescents' Snack Purchases
Status: Completed | Type: Observational
Sponsor: University at Buffalo (Other)
Responsible Party: Sarah-Jeanne Salvy, Ph.D., University at Buffalo
Other Study IDs: DB#2306
Record Dates: First submitted 2009-04-02; First posted 2009-04-03 (Estimated); Last update posted 2009-04-03 (Estimated); Status verified 2009-04

CONDITIONS: Social Influences; Food Consumption
Keywords: social influences; food purchases; childhood obesity; amount of energy dense food and beverage items purchased; amount of nutrient dense food and beverage items purchased
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to assess the effects of peer influences on snack purchases in adolescents. During the session teens will be given a certain amount of money to use to purchase foods and beverages in a hypothetical convenience store setting.

The investigators hypothesize that overweight youth will be less responsive to own-price elasticity for high calorie foods and less likely to show cross price elasticity for low calorie foods when the price of the high calorie for nutrient foods increases. The investigators also predict that overweight youth will show more cross price elasticity for low calorie foods when in the presence of peers; whereas lean youth's food purchases and price sensitivity will not be affected by the presence of peers.

ELIGIBILITY:
Inclusion Criteria:

* Boys and girls ages 12-14
* Youth must have at least a moderate liking of study foods used
* Youth must be at or above the 15th BMI percentile

Exclusion Criteria:

* Youth should have no dietary restrictions
* Youth should have no food allergies
* Youth should have no medical conditions that alter the body's ability to absorb nutrients or that can otherwise influence the participants' response to food

Ages: 12 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 2008-06; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah J Salvy, Ph.D., Principal Investigator — University at Buffalo
Locations (1):
- University at Buffalo, Division of Behavioral Medicine, Buffalo, New York, United States